CLINICAL TRIAL: NCT01157975
Title: A Randomized, Partially Blinded, Pilot Study of the Effects of Pioglitazone on HCV RNA in Overweight Subjects With Chronic HCV Genotypes 1 or 4 Infection.
Brief Title: Study the Relationship Between Obesity and Hepatitis C Replication
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was completed in another site
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Mario Chojkier, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 060913
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Pioglitazone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone (Experimental)
  Interventions: Drug: Pioglitazone
- Prednisone (Experimental)
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone will be taken at a dose of 30 mg for up to 14 days
  Other Names: ACTOS
  Arms: Pioglitazone
Drug: Prednisone — Prednisone will be taken at a dose of 40 mg for up to 4 days
  Arms: Prednisone

SUMMARY:
Patients with chronic hepatitis C viral infection (HCV) and with a BMI greater than 25Kg/m2 are refractory to medical treatment. Also, HCV replication seems to be affected when modeling insulin resistance in replicon cell culture systems.

PPARg -agonist (Pioglitazone) is effective in controlling liver inflammation in obese subjects with non-alcoholic steatohepatitis (NASH) and also improving insulin sensitivity. Therefore, we hypothesize that improving insulin resistance and /or inflammation may affect HCV replication and viral kinetics. Independently of PPARg pathways, Prednisone may increase HCV viral kinetics. .

DETAILED DESCRIPTION:
This is a randomized, two arm clinical trial. The investigators performing the primary and secondary endpoints are blinded to subject identifiers and arm identifiers.

Subject's screening for HCV Genotype 4 started in Agouza Hospital in July 2010 and ended in February, 2011. No recruitment has occurred for HCV Genotype 1.

ELIGIBILITY:
Inclusion Criteria:

* Infection with HCV genotype 1 or 4 (subjects infected with multiple genotypes are not eligible)
* BMI greater than 25 Kg/m2
* HCV-infected subjects naïve to treatment: subjects who either have never been treated for HCV infection or who previously received HCV treatment ending more than 3 months prior to enrollment for not longer than 2 weeks
* Plasma HCV RNA concentration of >10,000 IU/mL at the screening evaluation

Exclusion Criteria:

* Previous intolerance to Pioglitazone, Rosiglitazone, Troglitazone or corticosteroids
* Women who are pregnant or breastfeeding
* History of diabetes mellitus requiring treatment other than diet
* Decompensated liver disease or other known causes of liver disease including, but not limited to autoimmune hepatitis, Wilson's disease, hemochromatosis, primary biliary cirrhosis, schistosomiasis, sclerosing cholangitis, alcohol- or drug-induced liver disease, or alpha-one antitrypsin deficiency
* Concurrent hepatitis B virus (HBV) infection
* Known immunodeficiency disease, autoimmune disorders or active gastrointestinal disease
* Abuse of alcohol or illicit drugs within 6 months before enrollment
* Use of an investigational drug within 4 weeks before the screening visit or during the screening period.
* Use of systemic immunosuppressants
* History of poorly controlled psychiatric disease or poorly controlled pulmonary disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
HCV RNA | 2 weeks
  Only in the Pioglitazone group

SECONDARY OUTCOMES:
HCV RNA | Day 4
  Only in the Prednisone group
Serum indicators of insulin resistance (fasting glucose, insulin, lipids and serum retinol binding protein-4); adiponectins and inflammatory cytokines. | Day 14 (Pioglitazone) and Day 4 (Prednisone)
ALT and AST | Day 14 (Pioglitazone) and Day 4 (Prednisone)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Chojkier, MD, Principal Investigator — UCSD; Martina Buck, PhD, Principal Investigator — UCSD; Hesham Elkhayat, MD, Principal Investigator — Cairo University, Egypt
Locations (2):
- University of California at San Diego Hospitals, San Diego, California, United States
- Agouza Hospital, Giza, Egypt

REFERENCES:
- [Derived] Chojkier M, Elkhayat H, Sabry D, Donohue M, Buck M. Pioglitazone decreases hepatitis C viral load in overweight, treatment naive, genotype 4 infected-patients: a pilot study. PLoS One. 2012;7(3):e31516. doi: 10.1371/journal.pone.0031516. Epub 2012 Mar 7. PMID 22412837